CLINICAL TRIAL: NCT05598385
Title: Groin Complications in Open Vs. Percutaneous Peripheral Cannulation for Cardiopulmonary Bypass in Minimally Invasive Cardiac Surgery
Brief Title: Groin Complications in Open Vs. Percutaneous Peripheral Cannulation in Minimally Invasive Cardiac Surgery
Acronym: ProGlide-II
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: After the passing of the principal investigator, the clinical trial could not be started.
Sponsor: Jessa Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/148
Record Dates: First submitted 2022-10-26; First posted 2022-10-28 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
Keywords: Peripheral cannulation; Open cannulation; Percutaneous cannulation; Minimally invasive cardiac surgery
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Percutaneous cannulation (Active Comparator): Percutaneous peripheral cannulation will be applied. An ultrasound is performed preoperative, at discharge and during the follow-up consultation.
  Interventions: Procedure: Percutaneous cannulation
- Open cannulation (Active Comparator): Open peripheral cannulation will be applied. An ultrasound is performed preoperative, at discharge and during the follow-up consultation.
  Interventions: Procedure: Open cannulation

INTERVENTIONS:
Procedure: Open cannulation — A small incision is made to access the FA and FA. Afterwards, the incision site is traditionally closed with sutures.
  Arms: Open cannulation
Procedure: Percutaneous cannulation — Cannulation is performed through a suture-mediated closure system.
  Arms: Percutaneous cannulation

SUMMARY:
The aim of this randomized trial is to investigate the groin complications in open vs percutaneous peripheral cannulation for cardiopulmonary bypass in minimally invasive cardiac surgery

DETAILED DESCRIPTION:
The femoral artery (FA) and vein (FV) are considered the preferred site for peripheral cannulation during cardiac surgery. Normally, a small incision is made to access the FA and FV, which is also called open surgical cannulation. Afterwards, the incision site is traditionally closed with sutures (1, 2). However, groin complications such as hematoma, access-site infection and fistulas are complications that can eventually lead to a longer hospital stay (3).

Recently, suture-mediated closure systems (SMCS) have been developed to achieve hemostasis (4). This allows for percutaneous cannulation. Still, little is known about the effects on groin complications after percutaneous cannulation in cardiac surgery. Therefore, a prospective randomized study is now being conducted to investigate the groin complications in open vs. percutaneous peripheral cannulation for cardiopulmonary bypass in minimally invasive cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* >18 years
* Patients undergoing elective endoscopic cardiac surgery

Exclusion Criteria:

* Patients that do no understand Dutch, French, or English
* Heavily calcified cannula introduction site
* Central cannulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-11 (Estimated); Primary Completion 2024-11-09 (Actual); Study Completion 2024-11-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with groin complications | Until 30 days postoperatively
  Groin complications consist of groin-related bleeding, dissection, pseudoaneurysm, seroma, infection of the groin, artery occlusion, and reintervention in the groin. Groin complications are diagnosed by an ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Alaaddin Yilmaz, MD, Principal Investigator — Jessa Hospital

IPD SHARING:
Plan to Share IPD: No